CLINICAL TRIAL: NCT00906620
Title: Saving and Empowering Young Lives in Europe in Israel, Evaluation, Intervention and Prevention
Brief Title: Saving and Empowering Young Lives in Europe (Israel)
Acronym: SEYLE-ISRAEL
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, alan apter, Director of psychological medicine department at Schneider; Professor at Sackler School of medicine, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5277
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: Depression; Suicidality
Keywords: Data on student's healthy and at-risk lifestyles and their relation with health measured by well-being, depression and suicidality
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- QPR intervention (Experimental): QPR intervention (Question, Persuade & Refer): The QPR prevention program will be used in two modules, one for school staff and one for parents. According to the US Surgeon General's National Strategy for Suicide Prevention (2001), "key gatekeepers" are "people who regularly come into contact with individuals or families in distress" and gatekeeper training has been identified as one of a number of promising prevention strategies.
  Interventions: Other: QPR: question, persuade and refer (SEYLE)
- Awareness program (Experimental): The awareness programme is comprised of a leaflet, six posters and four seminars. The seminars are made up of one introductory lesson, and two interactive follow-up lessons with role play and one final meeting as a closing/debriefing lesson.
  Interventions: Other: QPR: question, persuade and refer (SEYLE)
- ProfScreen (Experimental): The program's primary objective is to help young people and their parents through the early identification of mental health problems, such as anxiety, depression, substance abuse, and suicide. Screening strategies are based on the valid premise that suicidal adolescents are under-identified, suffer from an active, often treatable mental illness such as depression and exhibit identifiable risk factors (Gould et al. 2003). A potential shortcoming of screening programs is that asking about suicide could increase suicidal ideation and behaviour. About this issue a recent study (Gould et al . 2005) on over 2300 students reported no evidence of iatrogenic effects of suicide screening and that screening in high schools is a safe component of youth suicide prevention efforts.
  Interventions: Other: QPR: question, persuade and refer (SEYLE)
- Control group (Experimental): The control group will comprise 250 subjects. After the baseline assessment, subjects will be randomized in one of the three intervention arms or in the control group. Individuals in the control group will undergo the same baseline and follow-up evaluations as subjects in the intervention arms and will receive the same leaflet about healthy lifestyles with information about the possibility to seek help for unhealthy, suicidal behaviour and mental health problems. In this arm, no additional intervention will be performed although the possibility of seeking help from mental health resources will be available.
  Interventions: Other: QPR: question, persuade and refer (SEYLE)

INTERVENTIONS:
Other: QPR: question, persuade and refer (SEYLE) — The QPR prevention program will be used in two modules, one for school staff and one for parents. According to the US Surgeon General's National Strategy for Suicide Prevention (2001), "key gatekeepers" are "people who regularly come into contact with individuals or families in distress" and gatekeeper training has been identified as one of a number of promising prevention strategies.

SUMMARY:
SEYLE is a health promoting program for adolescents in European schools. Its main objectives are to lead adolescents to better health through decreased risk-taking and suicidal behaviors, to evaluate outcomes of different preventive programs and to recommend effective culturally adjusted models for promoting health of adolescents in different European countries. Because of the significance of the SEYLE program and the importance of suicide research, Israel is honored to take part in this program and be a collaborator in it's implementation and research.

DETAILED DESCRIPTION:
In this health promotion program, a pilot intervention study will be implemented to assess the effects of three different health promoting / suicide prevention programs in 11,000 students across 11 European countries (Sweden, Austria, Estonia, France, Germany, Hungary, Ireland, Israel, Italy, Romania, Slovenia and Spain): 1. A general health promotion program targeting students' awareness on healthy/unhealthy behaviours and students' self-efficacy in diminishing unhealthy behaviours; 2. ProfScreen - screening by professionals of at-risk students through a questionnaire. For adolescents identified as high risk (screen positives) the program includes referral to mental health treatment and ensuring compliance. 3. QPR (Question, Persuade & Refer) - a gatekeepers' program, training all adult staff at schools (teachers, counselors, nurses etc.) and parents on how to recognize & refer a student with risk-taking behaviours or suffering from mental illness to mental-health help resources.

Each of these prevention programs uses a different active component in order to be successful. The first prevention program empowers the students by increasing their self-efficacy. The second prevention program (ProfScreen) empowers mental health professional in identifying subjects at risk. The third program (QPR) empowers teachers and parents in at-risk case finding and referring to mental health facilities. The registration of the complete RCT is available on the German Clinical Trials Registry (DRKS00000214).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between 13-17

Exclusion Criteria:

* none

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1247 (Actual)
Dates: Start 2009-09; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
evaluate the efficacy of different preventive programs. | 2012

SECONDARY OUTCOMES:
rate of risk taking behavior among adolescents | 2012

CONTACTS AND LOCATIONS:
Overall Officials: Alan Stanley Apter, MD, Principal Investigator — Schnider Children MC
Locations (1):
- Schnider Children MC, Petah Tikva, NON, Israel

REFERENCES:
- [Derived] Lustig S, Kaess M, Schnyder N, Michel C, Brunner R, Tubiana A, Kahn JP, Sarchiapone M, Hoven CW, Barzilay S, Apter A, Balazs J, Bobes J, Saiz PA, Cozman D, Cotter P, Kereszteny A, Podlogar T, Postuvan V, Varnik A, Resch F, Carli V, Wasserman D. The impact of school-based screening on service use in adolescents at risk for mental health problems and risk-behaviour. Eur Child Adolesc Psychiatry. 2023 Sep;32(9):1745-1754. doi: 10.1007/s00787-022-01990-z. Epub 2022 Apr 30. PMID 35488938
- [Derived] Carli V, Wasserman C, Wasserman D, Sarchiapone M, Apter A, Balazs J, Bobes J, Brunner R, Corcoran P, Cosman D, Guillemin F, Haring C, Kaess M, Kahn JP, Keeley H, Kereszteny A, Iosue M, Mars U, Musa G, Nemes B, Postuvan V, Reiter-Theil S, Saiz P, Varnik P, Varnik A, Hoven CW. The saving and empowering young lives in Europe (SEYLE) randomized controlled trial (RCT): methodological issues and participant characteristics. BMC Public Health. 2013 May 16;13:479. doi: 10.1186/1471-2458-13-479. PMID 23679917
- [Derived] Kelleher I, Keeley H, Corcoran P, Ramsay H, Wasserman C, Carli V, Sarchiapone M, Hoven C, Wasserman D, Cannon M. Childhood trauma and psychosis in a prospective cohort study: cause, effect, and directionality. Am J Psychiatry. 2013 Jul;170(7):734-41. doi: 10.1176/appi.ajp.2012.12091169. PMID 23599019